CLINICAL TRIAL: NCT02747108
Title: Improving Veteran Engagement in Diabetes Prevention (CDA 13-267)
Brief Title: ForgIng New Paths to Prevent DIabeTes (FINDIT)
Acronym: FINDIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Ann Arbor Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDX 15-001; CDA 13-267 (Other Grant/Funding Number: VA Health Services Research and Development)
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Prediabetes
Keywords: Veterans; Type 2 Diabetes Mellitus; Prediabetes; Decision-making; Motivation; Health Promotion; Prevention and Control
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood Test Group (Experimental): Patients will complete an HbA1c test and then receive brief counseling and written information about their test result based on the American Diabetes Association and National Diabetes Prevention Program guidelines.
  Interventions: Behavioral: Blood Test Group Intervention
- Brochure Group (usual care) (Active Comparator): Patients will not complete an HbA1c test and will instead receive brief counseling and written information about recommended screenings and immunizations.
  Interventions: Behavioral: Brochure Group Intervention

INTERVENTIONS:
Behavioral: Blood Test Group Intervention — Patients randomly assigned to the Blood Test Group will complete an HbA1c blood test around the time of their next primary care appointment. Following the HbA1c test, their VA primary care provider will be notified of the test result and will be provided with a detailed interpretation of the result. Trained study staff will then provide brief counseling by phone and written information by mail about their test result. The brief counseling and written information will be based on the American Diabetes Association and National Diabetes Prevention Program guidelines and will emphasize the risk of progression to type 2 diabetes mellitus and the rationale for preventive strategies, encourage aerobic exercise and a calorie-restricted diet to promote and maintain weight loss, and set a goal of achieving and sustaining a weight loss of at least 5% of body weight.
  Arms: Blood Test Group
Behavioral: Brochure Group Intervention — Participants will be asked to review a handout from the National Center for Health Promotion and Disease Prevention (NCP) on recommended screening tests and immunizations on or around the same date as their next primary care appointment.
  Arms: Brochure Group (usual care)

SUMMARY:
This study will evaluate the effects of screening for type 2 diabetes mellitus (T2DM) and brief counseling about screening test results on weight and key health behaviors among Veterans with risk factors for T2DM. Study participants will be randomly assigned to one of two study groups: (1) Blood Test Group or (2) Brochure Group. Participants in the Blood Test Group will complete a blood test called hemoglobin A1c (HbA1c) which measures average blood sugar levels. Participants will receive brief counseling about the results from their primary care provider or someone authorized to speak on their behalf. Participants randomly selected for the Brochure Group will review a handout from the VA National Center for Health Promotion and Disease Prevention (NCP) on recommended screening tests and immunizations. All participants will be asked to complete a survey prior to study group assignment, immediately after a Primary Care appointment, 3 months after enrollment, and 12 months after enrollment.

DETAILED DESCRIPTION:
An essential step in designing effective strategies to improve patient engagement in behavior change is to better understand their current levels of engagement in these behaviors and determine which factors most influence their engagement. Within and outside the Veterans Health Administration (VHA), little is known about how patients with risk factors for T2DM view their risk of developing T2DM, what these patients understand about strategies to reduce this risk, and to what degree at-risk patients are currently engaging in behaviors to prevent T2DM. This project will generate important new data in these areas and will improve the investigators' understanding of the effects of a prediabetes diagnosis and brief counseling on engagement in behaviors to prevent T2DM and mediators of these behaviors.

ELIGIBILITY:
Inclusion Criteria:

The investigators will recruit 315 non-diabetic Veterans receiving primary care at the Ann Arbor VA Medical Center who meet the following inclusion criteria:

* willing to complete a HIPAA authorization form
* no HbA1c results in previous 12 months
* due for VA Primary Care appointment approximately 12 weeks of sending a recruitment letter and who have a body-mass index (BMI) 30 kg/m2
* or BMI 25 kg/m2 with > 1 obesity-related condition such as:

  * hypertension
  * hyperlipidemia
  * Hypoalphalipoproteinemia
  * Coronary Artery Disease
  * Peripheral Vascular Disease
  * Hypertriglyceridemia
  * past hemoglobin A1c (HbA1c) of 5.7 - 6.4
  * past diagnosis of Impaired Fasting Glucose (IFG)
  * or Impaired Glucose Tolerance (IGT)
  * or Polycystic Ovary Syndrome (PCOS)

Exclusion Criteria:

* The investigators will exclude patients who are > 75 years of age
* are receiving chemotherapy for cancer, or have:

  * dementia
  * diabetes
  * dementia
  * New York Heart Association Class III or IV congestive heart failure
  * pregnancy
  * Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage 4 Chronic Obstructive Pulmonary Disease (COPD)
  * end-stage renal disease (ESRD)
  * cirrhosis
  * or have been hospitalized or received rehab for stroke or myocardial infarction within the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T. Kullgren, MD MPH MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kullgren JT, Youles B, Shetty S, Richardson C, Fagerlin A, Heisler M. ForgIng New paths in DIabetes PrevenTion (FINDIT): Study Protocol for a Randomized Controlled Trial. Trials. 2017 Apr 8;18(1):167. doi: 10.1186/s13063-017-1887-6. PMID 28388933

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans that met preliminary study eligibility criteria were mailed a letter about the study and were contacted by a Research Assistant 10 days later by phone to gauge their participation interest. Recruitment was conducted between December 2015 and February 2017.
Pre-assignment Details: Participants that met study criteria and had an upcoming primary care appointment were sent a Baseline Survey to complete as a requirement for randomization. Those that did not complete the Baseline Survey or whose primary care appointments were cancelled and not rescheduled were not randomized and thus excluded from analysis.
Groups:
- Blood Test Group: Patients will complete an HbA1c test and then receive brief counseling and written information about their test result based on the American Diabetes Association and National Diabetes Prevention Program guidelines.
  Blood Test Group Intervention: Patients randomly assigned to the Blood Test Group will complete an HbA1c blood test around the time of their next primary care appointment. Following the HbA1c test, their VA primary care provider will be notified of the test result and will be provided with a detailed interpretation of the result. Trained study staff will then provide brief counseling by phone and written information by mail about their test result. The brief counseling and written information will be based on the American Diabetes Association and National Diabetes Prevention Program guidelines and will emphasize the risk of progression to type 2 diabetes mellitus and the rationale for preventive strategies, encourage aerobic exercise and a calorie-restricted diet.
Period: Overall Study
Arm/Group | Blood Test Group | Brochure Group (Usual Care)
Started | 253 | 62
Completed | 248 | 60
Not Completed | 5 | 2
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants consist of Veterans randomized to either the Blood Test Group (Intervention Arm) and Brochure Group (Usual Care Arm).
Groups:
- Total: Total of all reporting groups
Arm/Group | Blood Test Group | Brochure Group (Usual Care) | Total
Number analyzed (Participants) | 253 | 62 | 315
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 133 | 32 | 165
  >=65 years | 120 | 30 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.01 (10.89) | 60.87 (11.83) | 60.98 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants randomized to each arm Population: The number of males and females randomized to each arm. Each column represents the arm whereas the row represents the gender with the row totaling the number of males and females that enrolled in the study.
  Participants
    Female | 22 | 5 | 27
    Male | 231 | 57 | 288
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 8
  Not Hispanic or Latino | 244 | 60 | 304
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 2 | 19
  White | 206 | 50 | 256
  More than one race | 23 | 2 | 25
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 253 | 62 | 315

OUTCOME MEASURES:

1. Primary Outcome: Weight Change From Baseline to 12 Months
Description: The primary outcome will be weight change 12 months after an HbA1c test and brief counseling or review of health promotion literature.
Time Frame: 12 months
Population: The population consisted of Veterans ages 75 and younger, who were due for an HbA1c lab, and met inclusion and exclusion criteria at the time of enrollment.
Measure: Mean (Standard Deviation); unit: Pounds
Groups:
- Blood Test Group (Normoglycemia): Participants in the Blood Test Group with Baseline HbA1c results in the normoglycemia range of less than 5.7.
- Blood Test Group (Prediabetes); Blood Test Group (Diabetes): Participants in the Blood Test Group with Baseline HbA1c results in the prediabetic range of 5.7 - 6.4.
Arm/Group | Blood Test Group (Normoglycemia) | Brochure Group (Usual Care) | Blood Test Group (Prediabetes) | Blood Test Group (Diabetes)
Number analyzed (Participants) | 112 | 54 | 90 | 10
Pounds | -.995535 (15.39902) | -2.1333341 (12.697408) | .039778 (12.69741) | -4.17 (9.906009)

2. Secondary Outcome: Change in Use of Medication for T2DM Prevention
Description: The investigators will use medical record data and survey data to evaluate changes in use of medication for T2DM prevention after an HbA1c test and brief counseling or review of health promotion literature.
Time Frame: 3 and 12 months
Population: The population consisted of veterans ages 75 and younger, who were due for an HbA1c lab, met inclusion and exclusion criteria at the time of enrollment, and had data available for this assessment
Measure: Count of Participants; unit: Participants
Groups:
- Blood Test Group (Prediabetes): Participants in the Blood Test Group with Baseline HbA1c results in the prediabetes range of n 5.7 - 6.4.
- Blood Test Group (Diabetes): Participants in the Blood Test Group with Baseline HbA1c results in the diabetes range of greater than 6.4.
Arm/Group | Blood Test Group (Normoglycemia) | Brochure Group (Usual Care) | Blood Test Group (Prediabetes) | Blood Test Group (Diabetes)
Number analyzed (Participants) | 134 | 62 | 106 | 11
Participants
  3 months: Metformin Use | 0 | 3 | 0 | 3
  3 months: No Metformin Use | 134 | 59 | 106 | 8
  12 months: Metformin Use | 2 | 3 | 2 | 2
  12 months: No Metformin Use | 132 | 59 | 104 | 9

3. Secondary Outcome: Changes in Participation in a Weight Management Program
Description: The investigators will use survey data to evaluate changes in participation in a weight management program after an HbA1c test and brief counseling or review of health promotion literature.
Time Frame: 3 months and 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Blood Test Group (Prediabetes): Participants in the Blood Test Group with Baseline HbA1c results in the prediabetes range of 5.7 - 6.4.
Arm/Group | Blood Test Group (Normoglycemia) | Brochure Group (Usual Care) | Blood Test Group (Prediabetes) | Blood Test Group (Diabetes)
Number analyzed (Participants) | 134 | 62 | 106 | 11
Participants
  3 months: Participated in weight management program | 17 | 8 | 8 | 2
  3 months: Did not participate in weight management program | 117 | 54 | 98 | 9
  12 months: Participated in weight management program | 20 | 10 | 8 | 2
  12 months: Did not participate in weight management program | 114 | 52 | 98 | 9

4. Secondary Outcome: Changes in Perception for Risk for T2DM
Description: The investigators will use survey data to evaluate changes in perception of risk for T2DM after an HbA1c test and brief counseling or review of health promotion literature. The Adriaanse T2DM Risk Perception Scale, which was included in the survey, measured self-assessed risk perception from 0 denoting no choice of developing T2DM to 100 denoting absolute confidence in developing T2DM.
Time Frame: Baseline, 2 weeks, 3 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- Blood Test Group (Prediabetes): Participants in the Blood Test Group with Baseline HbA1c results in the prediabetic range of 5.7 and 6.4.
- Blood Test Group (Diabetes): Participants in the Blood Test Group with Baseline HbA1c results in the diabetes range of 6.5 or higher.
Arm/Group | Blood Test Group (Normoglycemia) | Brochure Group (Usual Care) | Blood Test Group (Prediabetes) | Blood Test Group (Diabetes)
Number analyzed (Participants) | 134 | 63 | 107 | 11
Score on a scale
  Baseline | 20.775 (1.84) | 21.724 (2.611) | 27.596 (2.554) | 35.455 (6.112)
  2 weeks | 16.356 (1.704) | 23.684 (2.519) | 36.327 (2.41) | 56 (6.452)
  3 months | 19 (1.738) | 26.667 (3.036) | 35.851 (2.377) | 51.25 (6.031)
  12 months | 18.947 (1.943) | 23.585 (3.265) | 32.5 (2.504) | 43.333 (7.183)

5. Secondary Outcome: Changes in Knowledge of Strategies to Prevent T2DM
Description: The investigators will use survey data to evaluate changes in knowledge of strategies to prevent T2DM after an HbA1c test and brief counseling or review of health promotion literature. Respondents were given 3 open-ended questions to report things they could do to prevent T2DM. Each respective response to the 3 questions were coded and scored according to whether they indicated engagement in the following activities: weight loss, physical activity, use of metformin, or enrollment into a diabetes prevention program. Each question denoted with a positive response were coded with 1 whereas those that did not were coded as a 0. The three questions were summed into a final score ranging from 0 (no report of engagement in the aforementioned healthy activities) with the worst outcome to 3 (a report of 3 of the 4 aforementioned healthy activities) with the best outcome.
Time Frame: 2 weeks, 3 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Blood Test Group (Normoglycemia) | Brochure Group (Usual Care) | Blood Test Group (Prediabetes) | Blood Test Group (Diabetes)
Number analyzed (Participants) | 134 | 62 | 106 | 11
Score on a scale
  2 weeks | 1.03 (0.70) | 1.10 (0.65) | 1.34 (0.77) | 1.09 (0.70)
  3 months | 1.04 (0.64) | 1.01 (0.67) | 1.08 (0.66) | 1.09 (0.83)
  12 months | 1.03 (0.72) | 0.97 (0.68) | 1.08 (0.69) | 1.18 (0.87)

6. Secondary Outcome: Changes in Motivation to Prevent T2DM
Description: The investigators will use survey data to evaluate changes in motivation to prevent T2DM after an HbA1c test and brief counseling or review of health promotion literature. The Treatment Self-Regulation Questionnaire (TSRQ) was included in the survey and respondents were asked about their level of motivation from 1 (Not at all motivated) to 10 (Highly motivated).
Time Frame: Baseline, 2 weeks, 3 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Blood Test Group (Normoglycemia) | Brochure Group (Usual Care) | Blood Test Group (Prediabetes) | Blood Test Group (Diabetes)
Number analyzed (Participants) | 134 | 63 | 107 | 11
Score on a scale
  Baseline | 6.618 (.239) | 7.237 (.358) | 6.676 (.272) | 6.455 (.627)
  2 weeks | 6.558 (.24) | 7.246 (.321) | 7.67 (.215) | 7.9 (.432)
  3 months | 6.471 (.229) | 7.018 (.323) | 7.442 (.221) | 7 (.537)
  12 months | 6.793 (.234) | 6.981 (.371) | 7.207 (.236) | 6.889 (.897)

7. Secondary Outcome: Changes in Self-efficacy to Engage in Behaviors to Prevent T2DM
Description: The investigators will use survey data to evaluate changes in self-efficacy to engage in behaviors to prevent T2DM after an HbA1c test and brief counseling or review of health promotion literature. The Perceived Competence Scale was used to measure respondent self-efficacy from 1 (lowest) to 7 (highest).
Time Frame: Baseline, 3 months and 12 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Blood Test Group (Normoglycemia) | Brochure Group (Usual Care) | Blood Test Group (Prediabetes) | Blood Test Group (Diabetes)
Number analyzed (Participants) | 134 | 63 | 107 | 11
Score on a scale
  Baseline | 4.869 (.134) | 5.082 (.172) | 4.747 (.152) | 4.341 (.445)
  3 months | 4.926 (.125) | 5.005 (.192) | 4.826 (.148) | 4.906 (.432)
  12 months | 5.07 (.134) | 5.31 (.195) | 4.832 (.151) | 4.75 (.57)

8. Secondary Outcome: Change in Physical Activity
Description: The investigators will use survey data to evaluate changes in physical activity after an HbA1c test and brief counseling or review of health promotion literature. The International Physical Activity Questionnaire - Short Form (IPAQ-SF) was used to measure physical activity change. Respondents were asked to report how many hours and minutes within the past week they completed of vigorous physical activity, moderate physical activity, and brisk walking. The total sum of minutes for these three questions were subsequently coded into a yes/no binary variable for whether respondents met a recommended 150 minutes of overall physical activity within 7 days of being assessed. The values provided reflect a proportion of respondents that met or exceeded the 150 minute threshold of overall physical activity based on the newly generated variable that combined total minutes of vigorous physical activity, moderate physical activity, and brisk walking.
Time Frame: Baseline, 3 months and 12 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Proportion of Respondents
Arm/Group | Blood Test Group (Normoglycemia) | Brochure Group (Usual Care) | Blood Test Group (Prediabetes) | Blood Test Group (Diabetes)
Number analyzed (Participants) | 134 | 63 | 107 | 11
Proportion of Respondents
  Baseline | .542 (.044) | .5 (.066) | .495 (.047) | .273 (.138)
  3 months | .45 (.042) | .517 (.063) | .438 (.047) | .091 (.087)
  12 months | .489 (.043) | .5 (.063) | .457 (.047) | .364 (.145)

9. Secondary Outcome: Change in Mental Health
Description: The investigators will use survey data to evaluate changes in SF-12 mental health scores after an HbA1c test and brief counseling or review of health promotion literature. The SF-12 provides a calculation of (1) a physical score (PCS-12) generated from a subset of questions focused on physical health and (2) a mental health score (MCS-12) generated from a subset of questions focused on mental health. The data provided represent the mean score of the PCS-12 and MCS-12. Scores range from 0 to 100, where a zero score indicates the lowest level of physical/mental health measured by the scales and 100 indicates the highest level of physical/mental health.
Time Frame: Baseline, 2 weeks, 3 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Blood Test Group (Normoglycemia) | Brochure Group (Usual Care) | Blood Test Group (Prediabetes) | Blood Test Group (Diabetes)
Number analyzed (Participants) | 134 | 63 | 107 | 11
Score on a scale
  Baseline | 44.995 (9.63) | 44.264 (1.43) | 45.373 (1.086) | 37.926 (2.291)
  2 weeks | 46.366 (1.018) | 46.389 (1.496) | 46.512 (1.071) | 44.806 (2.548)
  3 months | 45.347 (1.037) | 48.249 (1.531) | 46.926 (1.095) | 48.703 (3.139)
  12 months | 47.082 (1.082) | 47.308 (1.37) | 47.58 (1.066) | 40.085 (4.352)

ADVERSE EVENTS:
Time Frame: Adverse events are reported for the full year of participation of each individual.
Description: Adverse events information was collected from participants if they reported events during phone correspondence with a Research Assistant related to the brief intervention, 2-week, 3-month, and 12-month surveys.
Arm/Group | Blood Test Group | Brochure Group (Usual Care)
All-Cause Mortality (participants affected / at risk) | 2/253 | 2/62
Serious Adverse Events (participants affected / at risk) | 0/253 | 0/62
Other Adverse Events (participants affected / at risk) | 3/253 | 1/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blood Test Group (N=253) | Brochure Group (Usual Care) (N=62)
Surgical and medical procedures (Surgical and medical procedures) | 2 (2) | 0 (0)
Self-report of cold/flu/sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diagnosis of cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Serious depression (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT02747108/Prot_SAP_000.pdf